CLINICAL TRIAL: NCT02319707
Title: Management of the Third Stage of Labor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yariv yogev (Other)
Responsible Party: Sponsor-Investigator, Yariv yogev, Prof. Yariv Yogev Director, Division of obstetrics and delivery, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0553-14-RMC
Record Dates: First submitted 2014-12-14; First posted 2014-12-18 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intramuscular treatment:IV (Experimental): pregnant women, 34-41 weeks of gestation, which were treated with 10 IU of IM Oxytocin during the third stage of labor.
  Interventions: Drug: Oxytocin
- Combined treatment:IV+IM (Experimental): pregnant women, 34-41 weeks of gestation, which were treated with 10 IU of IM Oxytocin together with 10 IU of IV Oxytocin in 100 ml NaCl 0.9% during the third stage of labor.
  Interventions: Drug: Oxytocin
- The control group (Active Comparator): pregnant women, 34-41 weeks of gestation, which were treated with 10 IU of IV Oxytocin in 100 ml NaCl 0.9% during the third stage of labor. (this is the routine practice in our department).
  Interventions: Drug: Oxytocin in 100 ml NaCl 0.9%

INTERVENTIONS:
Drug: Oxytocin — The study group: divided into two groups:
  • Intramuscular treatment: pregnant women, 34-41 weeks of gestation, which were treated with 10 IU of IM Oxytocin during the third stage of labor.
  • Combined treatment: pregnant women, 34-41 weeks of gestation, which were treated with 10 IU of IM Oxytocin together with 10 IU of IV Oxytocin in 100 ml NaCl 0.9% during the third stage of labor.
  Other Names: Pitocin
  Arms: Combined treatment:IV+IM; Intramuscular treatment:IV
Drug: Oxytocin in 100 ml NaCl 0.9% — The control group:
  pregnant women, 34-41 weeks of gestation, which were treated with 10 IU of IV Oxytocin in 100 ml NaCl 0.9% during the third stage of labor. (this is the routine practice in our department).
  Arms: The control group

SUMMARY:
To compare the efficacy of three different protocols of third stage management in preventing PPH.

DETAILED DESCRIPTION:
The third stage of labor refers to the period following the completed delivery of the newborn until the completed delivery of the placenta. The length of the third stage and its complications are affected by the uterine contractility and the duration of placental separation. The normal duration of third stage in nulliparous as well as in multiparous women is less than 30 minutes. There is strong evidence supporting the routine administration of uterotonic agents for the prevention of post-partum hemorrhage (PPH), in order to enhance natural uterine contraction in the third stage of labor, thus reducing the occurrence of PPH by 40%.

There is a joint policy statement between the International Confederation of Midwives (ICM), the International Federation of Gynecology and Obstetrics (FIGO) and the World Health Organization (WHO), all of which recommend active management of the third stage of labor in order to prevent PPH. active management led to a reduction in PPH incidence, maternal Hemoglobin<9g/dL and need for blood transfusion. (4-7).

Active management of the third stage of labor involves prophylactic uterotonic treatment, early cord clamping and controlled cord traction to deliver the placenta. (2) Oxytocin is the first agent of choice for PPH prophylaxis because of its high efficacy and a low incidence of associated side effects. (6-9). Cotter et al found that the use of Oxytocin for PPH prophylaxis in the third stage of labor decreased the rate of maternal blood loss greater than 500 ml by approximately 50%. (10).

Oxytocin route of administration is either intravenously (IV) or intramuscularly (IM), with no significant difference in PPH incidence (9). This is based on a pharmacokinetic research from 1972 which found no difference between the absorption rates in both routes of administration. Since then no further research targeting this question was preformed. (11-12). recent guidelines from WHO, FIGO and ICM all recommended the use of 10 IU Oxytocin IM. (4, 7,13).

Previous studies have investigated the effect of intra-umbilical vein Oxytocin injection in reducing blood loss during the third stage of labor. This route of administration directs treatment to the placental bed and uterine wall, resulting in earlier uterine contraction and placental separation. However, limited published literature is available evaluating the effect of umbilical vein oxytocin injection in routine practices for active management of the third stage of labor. A prospective, randomized controlled trial of 412 women found that intra-umbilical injection of oxytocin alongside active management of the third stage of labor significantly reduced postpartum blood loss and the duration of the third stage (14).

Other uterotonic agents including Syntometrine (IM), Ergometrine (IM or IV) and Misoprostol (IM), can be used in active management of the third stage of labor. However, high quality evidence regarding their efficacy compared to Oxytocin is scarce. (9-10)

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* 34-41 weeks of gestation.
* Maternal age between 18 and 45.

Exclusion Criteria:

* Women who enter delivery room during the active phase of labor (cervical dilatation greater than 5 cm)
* Coagulation defects
* VAS score>3 (pain score)
* Women with early PPH
* Suspected placental abruption

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin concentration during labor | first and second day after delivery

SECONDARY OUTCOMES:
Blood count (CBC) on the first and second day after delivery | first and second day after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Yariv Yogev, professor, Principal Investigator — Director, Division of obstetrics and delivery

REFERENCES:
- [Derived] Oladapo OT, Okusanya BO, Abalos E, Gallos ID, Papadopoulou A. Intravenous versus intramuscular prophylactic oxytocin for the third stage of labour. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD009332. doi: 10.1002/14651858.CD009332.pub4. PMID 33169839